CLINICAL TRIAL: NCT07392216
Title: Functional Ovarian Reserve in Sickle Cell Disease
Status: Not yet recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FORSCD
Record Dates: First submitted 2026-01-26; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Disease
Keywords: Ovary Function; Sickle Cell Disease; Children; Female; Puberty; Anti-Mullerian Hormone (AMH); Healthy Controls
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Sickle Cell Disease: Females with sickle cell disease, all genotypes (age at enrollment ≥ 10 years and < 19 years)
- Healthy Controls: Healthy female siblings/relatives of patients with SCD (including those with sickle cell trait), and other females of similar race/ethnicity (age at enrollment ≥ 10 years and < 19 years)

SUMMARY:
This study aims to look at AMH levels in female children with SCD as they go through puberty to see if they are at the same level as other children without SCD at the same age and/or pubertal stage and will also look at how treatment exposures and pain crises affect the AMH levels in children with SCD.

Primary Objective:

* To evaluate whether AMH levels are lower in pre-teens and adolescent females with SCD when compared with healthy female controls (siblings, relatives, non-relatives of similar race/ethnicity) at the same age and pubertal stage.

Secondary Objectives:

* To evaluate whether AMH has a similar trajectory in female pre-teens and adolescents with SCD when compared with the general population and controls.
* To describe pubertal timing, menstrual history, and markers of functional ovarian reserve (FOR), as well as prevalence of premature ovarian insufficiency (POI) as determined by medical history and laboratory markers in pre-teens and adolescents with SCD in comparison with their female controls.
* To correlate AMH levels with FSH and estradiol levels, normal pubertal timing, and menstrual history in children and adolescents with SCD.
* To correlate the severity of SCD (number of vaso-occlusive events) with pubertal timing, presence of normal vs abnormal menstruation, and laboratory markers of FOR, in pre-teens and adolescents with SCD.
* To correlate the use of SCD modifying treatment modalities with pubertal timing, menstrual pattern, and laboratory markers of FOR in pre-teens and adolescents with SCD.

DETAILED DESCRIPTION:
This is a non-therapeutic cross-sectional two-year pilot study within an eight-year longitudinal study.

After the parent and/or patient has given permission to enroll on the research study, review of the electronic medical record and SCCRIP (NCT02098863) data base will be performed to obtain data on current medical therapy, number of vaso-occlusive events and types of events as well as ED or hospital visits, laboratory studies and use of sickle cell disease modifying therapies.

A questionnaire will be distributed annually from time of enrollment until age 19.0 years to participants with SCD and consenting legal guardian (if applicable). For healthy controls, the same questionnaire will be provided to coincide with their one-time research visit. Pubertal status will be collected from questionnaires (prepubertal/no breast tissue, pubertal (breast tissue, but no menses), post-menarcheal. For those menstruating, regularity of menses will be ascertained through questionnaire answers and also date of last menstrual period. Questions for participants will also include questions regarding all forms of hormonal contraception and current opiate-containing medications.

For subjects with SCD, blood will be collected at the time of a clinic visit and occur concurrently with an already scheduled lab draw for clinical care with a goal frequency of annually. For controls, blood will be collected at a one-time study visit.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease of any genotype or a healthy sibling, relative, household member, or other females of similar race/ethnicity of a patient with sickle cell disease
* Age at enrollment ≥ 10 years and < 19 years
* Females

Exclusion Criteria:

* History of hematopoietic stem cell transplantation or gene therapy prior to enrollment or preparing for hematopoietic stem cell transplantation or gene therapy prior to enrollment
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent
* Pregnancy

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Females with Sickle cell disease of any genotype or a healthy sibling, relative, household member, or other females of similar race/ethnicity of a patient with sickle cell disease
Study Population: Females with Sickle cell disease of any genotype or a healthy sibling, relative, household member, or other females of similar race/ethnicity of a patient with sickle cell disease
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
Difference in AMH levels in pre-teens and adolescent females with SCD compared with healthy female controls (siblings, relatives, or non-relatives) at the same age | Earliest AMH collection after enrollment, up to 2 years after study activation
  Investigators will address this by targeting the relative difference in mean. For each participant, the earliest AMH measurement will be used. All patients recruited during the cross-sectional stage with at least 1 AMH measurement will be evaluable for the analysis, except for patients who have received hematopoietic stem cell transplant (HSCT) or gene therapy before their first study AMH measurement. Patients who either (1) have no available AMH at the end of the cross-sectional phase or (2) received HSCT or gene therapy before their first study AMH measurement will be considered unevaluable for this analysis.
Difference in AMH levels in pre-teens and adolescent females with SCD compared with healthy female controls (siblings, relatives, or non-relatives) at the same pubertal stage | Earliest AMH collection after enrollment, up to 2 years after study activation
  Investigators will address this by targeting the relative difference in mean. For each participant, the earliest AMH measurement will be used. Pubertal status will be defined as a nominal variable with the following categories: prepubertal, pubertal but premenarchal, postmenarchal, and 3 years postmenarchal. This will be derived from the self-reported status of any breast development and experiencing menarche by the time of the visit with the AMH draw.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Yu, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols